

Protocol 1936-201-008 Amd 1

# Title Page

**Protocol Title**: A Phase 2 Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety and Efficacy of BOTOX® (Botulinum Toxin Type A) Purified Neurotoxin Complex for the Treatment of Platysma Prominence

**Protocol Number**: 1936-201-008

Amendment Number: Amendment 1

Product: BOTOX® (botulinum toxin type A) purified neurotoxin complex (United States and

Canada adopted name is onabotulinumtoxinA)

**Brief Protocol Title**: BOTOX for the Treatment of Platysma Prominence

**Development Phase:** Phase 2

#### Sponsor Name and Legal Registered Address:

Allergan Sales LLC Allergan Limited

5 Giralda Farms 1st Floor Marlow International, The Parkway

Madison, NJ 07940 Marlow, Buckinghamshire, SL7 1YL

USA UK

Regulatory Agency Identifying Number(s): IND 133,036

**Emergency Telephone Number** Refer to the study contacts page

#### SAE Reporting Fax Number/Email:

IR-CLINICAL-SAE@Allergan.com Fax +1-714-796-9504 or Back-up Fax +1-714-246-5295

#### **Sponsor Signatory**:



Refer to the final page of this protocol for electronic signature and date of approval.



# **Protocol Amendment Summary of Changes Table**

| DOCUMENT HISTORY | |
|-------------------|---------------|
| Document | Date |
| Amendment 1 | August 2019 |
| Original Protocol | February 2019 |

#### Amendment 1 (August 2019)

#### Overall Rationale for the Amendment:

The overall rationale for the changes implemented in Protocol Amendment 1 was to make the eligibility criteria less restrictive





# **Table of Contents**

| | age | |
|---|---|---|
| | of Contents | |
| | Tables | |
| | Figures | |
| 1. | Protocol Summary | 7 |
| 1.1.<br>1.2. | Synopsis | |
| 2. | Introduction | 12 |
| 2.1. | Study Rationale | |
| <ul><li>2.2.</li><li>2.3.</li></ul> | Background Benefit/Risk Assessment | |
| 3. | Objectives and Endpoints | |
| 4. | Study Design | |
| 4.1.<br>4.2. | Overall Design | |
| 4.3. | Justification for Dose | |
| 4.4. | End of Study Definition | |
| 5. | Study Population | 20 |
| 5.1. | Inclusion Criteria | |
| 5.2. | Exclusion Criteria | |
| 5.3.<br>5.4. | Lifestyle Considerations | |
| | Screen Failures | |
| <b>6.</b> 6.1. | Study Intervention | |
| 6.2. | Preparation/Handling/Storage/Accountability | |
| 6.3. | Measures to Minimize Bias: Randomization and Blinding | |
| 6.4. | Study Intervention Compliance | 29 |
| 6.5. | Concomitant Therapy | |
| 6.5.1. | Prohibited Interventions and Washout Before the Study | |
| 6.5.2.<br>6.5.3. | Permitted Interventions | |
| 6.6. | Dose Modification | |
| 6.7. | Intervention after the End of the Study | |
| 7. | Discontinuation of Study Intervention and Participant | |
| | Discontinuation/Withdrawal | 30 |



# BOTOX

| 7.1. | Discontinuation of Study Intervention | 3 |
|---------|--------------------------------------------------------------|----|
| 7.2. | Participant Discontinuation/Withdrawal from the Study | |
| 7.3. | Lost to Follow Up | |
| 8. | Study Assessments and Procedures | 32 |
| 8.1. | Efficacy Assessments | |
| 8.1.1. | Primary Efficacy Assessment | |
| 8.1.2. | Secondary Efficacy Assessment | |
| 8.1.3. | Exploratory Efficacy Assessments | |
| 8.2. | Safety Assessments | |
| 8.2.1. | Height and Weight | |
| 8.2.2. | Vital Signs | |
| 8.2.3. | Pregnancy Testing | |
| 8.3. | Adverse Events and Serious Adverse Events | |
| 8.3.1. | Time Period and Frequency for Collecting Adverse Event and | |
| | Serious Adverse Event Information | 3 |
| 8.3.2. | Method of Detecting Adverse Events and Serious Adverse | |
| 0.0.2. | Events | 3′ |
| 8.3.3. | Follow-up of Adverse Events and Serious Adverse Events | |
| 8.3.4. | Regulatory Reporting Requirements for Serious Adverse Events | |
| 8.3.5. | Pregnancy | |
| 8.3.7. | Medication Errors | 30 |
| 8.4. | Treatment of Overdose | |
| 8.5. | Pharmacokinetics | |
| 8.6. | Pharmacodynamics | |
| 8.7. | Genetics | |
| 8.8. | Biomarkers and Other Assessments | |
| 8.9. | Health Economics | |
| 9. | Statistical Considerations | |
| 9.1. | Statistical Hypotheses | |
| 9.2. | Sample Size Determination | |
| 9.3. | Populations for Analyses | |
| 9.4. | Statistical Analyses | |
| 9.4.1. | Efficacy Analyses | |
| 9.4.2. | Safety Analyses | |
| 9.4.3. | Other Analyses | |
| 9.5. | Interim Analyses | 44 |
| 10. | Supporting Documentation and Operational Considerations | 4 |
| 10.1. | Appendix 1: Regulatory, Ethical, and Study Oversight | |
| | Considerations | 45 |
| 10.1.1. | Regulatory and Ethical Considerations | |
| 10.1.2. | Financial Disclosure. | |



Table 6-2

Table 8-1

Table 8-2

| BOTOX | | |
|----------|------------------------------------------------------------|----|
| 10.1.3. | Informed Consent Process | 46 |
| 10.1.4. | Data Protection. | 46 |
| 10.1.5. | Posting Clinical Study Data | 46 |
| 10.1.6. | Data Quality Assurance | 47 |
| 10.1.7. | Source Documents | 47 |
| 10.1.8. | Study and Site Closure | 48 |
| 10.1.9. | Publication Policy | 48 |
| 10.1.10. | Compliance with Protocol. | |
| 10.2. | Appendix 2: Clinical Laboratory Tests | 50 |
| 10.3. | Appendix 3: Adverse Events: Definitions and Procedures for | |
| | Recording, Evaluating, Follow-up, and Reporting | 51 |
| 10.4. | Appendix 4: Abbreviations | |
| 10.5. | Appendix 5: Standard Discontinuation Criteria | |
| 10.6. | Appendix 6: Study Tabular Summary | 59 |
| 10.7. | Appendix 7: Contraceptive Guidance and Collection of | |
| | Pregnancy Information | |
| 10.8. | Appendix 8: Clinician Allergan Platysma Prominence Scale . | |
| 10.9. | Appendix 9: Participant Allergan Platysma Prominence Scale | 65 |
| 11. | References | 86 |
| | List of Tables | |
| Table 6- | Number of Injection and Total Dose | 26 |
| Table 0- | i italioti of injection and Total Dosc | |

# 

Clinician Allergan Platysma Prominence Scale (C-APPS) at Maximum



| Protocol 1936-201-008 Amd 1 |
|-----------------------------|
| 42 |
| ds62 |
| of the Platysma Muscle |
| 14 |
| of |



## 1. Protocol Summary

## 1.1. Synopsis

**Protocol Title**: A Phase 2 Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety and Efficacy of BOTOX® (Botulinum Toxin Type A) Purified Neurotoxin Complex for the Treatment of Platysma Prominence

**Protocol Number:** 1936-201-008

Amendment Number: Amendment 1

Brief Title: BOTOX for the Treatment of Platysma Prominence

Study Rationale:



BOTOX treatment is expected to improve the appearance of platysma prominence by minimizing the visible effects of platysma muscle contraction. The purpose of this placebocontrolled Phase 2 trial is to evaluate the safety and efficacy of a high and a low dose of BOTOX compared with placebo to reduce the appearance of platysma prominence in adult participants with moderate to severe platysma prominence.

Objectives and Endpoints:

| Objectives | Endpoints |
|---|---|
| Primary | Primary |
| To evaluate the efficacy of a high and low dose of BOTOX compared with placebo in participants with moderate to severe platysma prominence at maximum contraction, as rated by the investigator To evaluate the safety of a high and low dose of BOTOX compared with placebo in participants with moderate to severe platysma prominence | Achievement of at least a 1-grade improvement at Day 14, as rated at maximum contraction by investigator using the Clinician Allergan Platysma Prominence Scale (C-APPS) Incidence of adverse events and changes from baseline in vital signs |
| Secondary | Secondary |
| To evaluate the efficacy of a high and low dose of<br>BOTOX compared with placebo in participants with<br>moderate to severe platysma prominence at<br>maximum contraction, as rated by the participant | Achievement of at least a 1-grade improvement at Day 14, as rated at maximum contraction by participant using the Participant Allergan Platysma Prominence Scale (P-APPS) |



#### BOTOX

| Objectives | Endpoints |
|-------------|-------------|
| Exploratory | Exploratory |

#### **Overall Study Design:**

This is a 4-month, multicenter, randomized, double-blind, placebo-controlled, dose-ranging study to assess the efficacy and safety of single-treatment BOTOX in adult participants with moderate to severe platysma prominence. After verification that the participants have met all inclusion and exclusion criteria, and have completed all baseline study procedures, participants will be randomized in a 1:1:1 ratio to receive BOTOX high dose, BOTOX low dose, or placebo.

There are 8 scheduled study visits: screening (Day -14 to Day -7), randomization/study intervention (Day 1), follow-up visits (Days 7, 14, 30, 60, and 90), and study exit (Day 120).

#### **Number of Participants:**

Approximately 165 participants will be enrolled. Based on an anticipated dropout rate of 10%, 148 participants will be analyzable for the primary endpoint.

#### **Number of Sites:**

Approximately 15 sites in the United States and Canada

#### **Intervention Groups and Study Duration:**

Study participants will be randomized in a 1:1:1 allocation ratio to receive BOTOX high dose, BOTOX low dose, or placebo.

The highest possible total

dose to be administered to a participant is U.





The total study duration is approximately 4 months.

Data Monitoring Committee: Not applicable



# 1.2. Schedule of Activities (SoA)

Procedures are recommended to be done in sequence as listed in the schedule below, unless otherwise stated.

| | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visits 7 | Visit 8 |
|---|---|---|---|---|---|---|---|---|
| Study Procedures | Screening<br>Day -14<br>to Day -7 | Baseline/<br>Randomization/<br>Intervention<br>Day 1 <sup>a</sup> | Day 7 | Day 14 | Day 30 | Day 60 | Day 90 | Study<br>Exit <sup>b</sup><br>Day 120 |
| Visit Windows | - | - | ± 3 Days | ± 3 Days | ± 3 Days | ± 7 Days | ± 7 Days | ± 7 Days |
| Informed Consent, Privacy Authorization | X | | | | | | | |
| Inclusion/Exclusion Criteria | X | X | | | | | | |
| Demographics | X | | | | | | | |
| Medical/Surgical History | X | | | | | | | |
| Weight | X | X | X | X | X | X | X | X |
| Fitzpatrick Skin Phototype <sup>d</sup> | X | | | | | | | |
| Abbreviated Physical Examination <sup>e</sup> | X | | | | | | | |
| Vital Signs <sup>f</sup> | X | X | X | X | X | X | X | X |
| Urine Pregnancy Test (WOCBP only) <sup>g</sup> | X | X | | | | | | X |
| Standardized Photography | X | X | X | X | X | X | X | X |
| Self-Assessment by Participants: | | | | | | | | |
| Participant Allergan Platysma Prominence Scale (P-APPS) <sup>i</sup> | | X | X | X | X | X | X | X |



#### **BOTOX**

| | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visits 7 | Visit 8 |
|---|---|---|---|---|---|---|---|---|
| Study Procedures | Screening<br>Day -14<br>to Day -7 | Baseline/<br>Randomization/<br>Intervention<br>Day 1 <sup>a</sup> | Day 7 | Day 14 | Day 30 | Day 60 | Day 90 | Study<br>Exit <sup>b</sup><br>Day 120 |
| Visit Windows | - | - | ± 3 Days | ± 3 Days | ± 3 Days | ± 7 Days | ± 7 Days | ± 7 Days |
| Clinician Assessment: | | | | | | | | |
| Clinician Allergan Platysma Prominence Scale (C-APPS) | X | X | X | X | X | X | X | X |
| Randomization | | X | | | | | | |
| Study Intervention Administration <sup>j</sup> | | X | | | | | | |
| Concomitant Medications/Procedures | X | X | X | X | X | X | X | X |
| Adverse Events <sup>k</sup> | X | X | X | X | X | X | X | X |

All baseline (Day 1) study procedures, including patient-reported outcome questionnaires, must be completed before randomization and study intervention.

Or early discontinuation from the study. All exit assessments should be completed as soon as possible after a decision to discontinue a participant from the study. c

Fitzpatrick Skin Phototype is provided in Section 10.11.

An abbreviated physical examination will be completed at the screening visit and will include the investigator assessment of general appearance, head, ears, eyes, nose, throat (HEENT), and

Vital Signs (blood pressure, respiratory rate, pulse rate) will be taken while the participant is sitting for at least 5 minutes.

Woman of childbearing potential (WOCBP) must have a negative urine test result before receiving study intervention. A urine pregnancy test may also be performed at any other visit, at the investigator's discretion.

Prepared by an Independent Drug Reconstitutor (IDR) and injected by the investigator. NOTE: The IDR must not perform any other study-related procedures.

On Day 1, AEs will be collected prior to and after treatment. Participants will be observed at least 30 minutes after study intervention administration for AEs. In the case of an AESI, see Section 8.3.6.

d



#### 2. Introduction

Botulinum toxin type A purified neurotoxin (BOTOX®) is approved to treat a variety of medical conditions and was first approved for therapeutic treatment of facial spasmodic disorders in 1989. BOTOX was first approved for aesthetic treatment of glabellar lines in 2002, and today is one of the most popular nonsurgical procedures in aesthetic medicine (ASAPS 2017 Cosmetic Surgery National Data Bank Statistics). When BOTOX is injected into a muscle, it interferes with neuromuscular transmission, producing a temporary chemical denervation resulting in localized relaxation of the muscle and reduction in muscle activity. In the upper face, BOTOX treatment improves the appearance of lines (wrinkles on the skin surface) associated with repeated muscle activity.

BOTOX may be a preferred treatment alternative to cosmetic surgery because its effects are temporary, less invasive with the potential for fewer serious side effects, and not anticipated to require a long recovery time, while producing a relatively rapid, predictable, and desired effect on platysma muscle activity.

A detailed description of the safety and efficacy experience of BOTOX is provided in the IB.

## 2.1. Study Rationale

BOTOX treatment is expected to improve the appearance of platysma prominence associated by minimizing the visible effects of platysma muscle contraction.

The purpose of this placebo-controlled Phase 2 trial is to evaluate the safety and efficacy of a high and a low dose of BOTOX compared with placebo to reduce the appearance of platysma prominence in adult participants with moderate to severe platysma prominence.







BOTOX



Figure 2-1 The Platysma Muscle: Anterior and Posterior Margins of the Platysma Muscle Sheets



Source: Grant's Atlas of Anatomy, 14th Edition

# 2.3. Benefit/Risk Assessment







More detailed information about the expected benefits and risks and reasonably expected AEs of BOTOX may be found in the IB.



# 3. Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary | Primary |
| To evaluate the efficacy of a high and low dose of BOTOX compared with placebo in participants with moderate to severe platysma prominence at maximum contraction, as rated by the investigator To evaluate the safety of a high and low dose of BOTOX compared with placebo in participants with moderate to severe platysma prominence | Achievement of at least a 1-grade improvement at Day 14, as rated at maximum contraction by investigator using the Clinician Allergan Platysma Prominence Scale (C-APPS) Incidence of adverse events and changes from baseline in vital signs |
| Secondary | Secondary |
| To evaluate the efficacy of a high and low dose of<br>BOTOX compared with placebo in participants with<br>moderate to severe platysma prominence at<br>maximum contraction, as rated by the participant | Achievement of at least a 1-grade improvement at Day 14, as rated at maximum contraction by participant using the Participant Allergan Platysma Prominence Scale (P-APPS) |
| Exploratory | Exploratory |



### 4. Study Design

#### 4.1. Overall Design

This is a 4-month, multicenter, randomized, double-blind, placebo-controlled, dose-ranging study with approximately 165 enrolled participants to assess the efficacy and safety of single-treatment BOTOX in adult participants with moderate to severe platysma prominence. The study will be conducted in the United States and Canada at approximately 15 study sites.

After verification that the participant meets all inclusion and exclusion criteria, and completion of all baseline study procedures, they will be randomized on Day 1. Study participants will be randomized in a 1:1:1 allocation ratio to receive BOTOX high dose, BOTOX low dose, or placebo.

There are 8 scheduled study visits: screening (Day -14 to Day -7), randomization/study intervention (Day 1), follow-up visits (Days 7, 14, 30, 60, and 90), and study exit (Day 120).

Approximately 165 participants will be enrolled. Based on an anticipated dropout rate of 10%, 148 participants will be analyzable for the primary endpoint.

## 4.2. Scientific Rationale for Study Design

Clinical experience and literature sources suggest that the use of botulinum toxin type A has beneficial effects on platysma prominence. Using a rigorous study design that is randomized, double-blind, and placebo-controlled, this study will provide information regarding the safety and efficacy of BOTOX versus placebo for the treatment of platysma prominence.

The sponsor developed the C-APPS as a clinician's assessment tool for evaluation of platysma prominence at maximum contraction. In the present study, all investigators will be trained to properly use the C-APPS to evaluate and grade the severity of platysma prominence at maximum contraction

The P-APPS has been developed as a participant self-assessment tool for evaluation of platysma prominence at maximum contraction.





# 4.3. Justification for Dose







This dose ranging study will evaluate the efficacy and safety of single-treatment BOTOX in adult participants with moderate to severe platysma prominence. Study participants will be randomized in a 1:1:1 allocation ratio to receive BOTOX high dose, BOTOX low dose, or placebo, and study participants could receive up to U of BOTOX in this study (Section 6.1).

# 4.4. End of Study Definition

The End of Study (EOS) Visit is defined as the date of the last visit of the last participant.

A participant is considered to have completed the study if he/she has completed all phases of the study including the last visit.



# 5. Study Population



Prospective approval of protocol deviations to recruitment and enrollment criteria, also known as protocol waivers or exemptions, is not permitted.

## 5.1. Inclusion Criteria

Participants are eligible to be included in the study only if all the following criteria apply:

| 1. | Age |
|---|---|
| 1.01 | Participant must be at least 18 years of age (or older if legal age of adulthood is > 18 per local regulations) at the time of signing the informed consent |
| 2. | Type of Participant |
| 2.01 | Participants must have the ability to correctly and maximally contract their platysma muscle |
| 2.02 | |
| 2.03 | |
| 3. | Weight and Body Mass Index |
| 3.01 | |
| 4. | Sex |
| 4.01 | Male or female |



#### **BOTOX**

| 5. | Contraceptives |
|---|---|
| 5.01 | Female participants willing to minimize the risk of inducing pregnancy for the duration of the clinical study and follow-up period |
| 5.02 | A female participant is eligible to participate if she is not pregnant (has a negative urine pregnancy result prior to randomization; see Appendix 7), not breastfeeding, and at least one of the following conditions applies: |
| | <ul> <li>a. Not a woman of childbearing potential (WOCBP) as defined in Appendix 7 OR</li> <li>b. A WOCBP who agrees to follow the contraceptive guidance in Appendix 7 during the treatment and follow-up period through study exit.</li> </ul> |
| 6. | Informed Consent |
| 6.01 | Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol |
| 6.02 | Written informed consent from the participant has been obtained prior to any study-related procedures |
| 6.03 | Written documentation has been obtained in accordance with the relevant country and local privacy requirements, where applicable |
| 7. | Other |
| 7.01 | Able, as assessed by the investigator, and willing to read and follow study instructions and likely to complete all study assessments and required study visits |

# 5.2. Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

| 1. | Medical Conditions |
|------|--------------------|
| 1.01 | |



#### **BOTOX**









#### BOTOX

| 4.05 | History of alcohol or drug abuse within 12 months of the study |
|---|---|
| 4.08 | Directly or indirectly involved in the conduct and administration of this study as an investigator, subinvestigator, study coordinator, or other study staff member; or employee of the sponsor or a first-degree family member, significant other, or relative residing with one of the above persons involved directly or indirectly in the study; or enrolled in the study at another clinical site |

#### 5.3. Lifestyle Considerations

#### 5.4. Screen Failures

Screen failures are defined as participants who consent to participate in the clinical study but are not subsequently randomly assigned to study intervention/entered in the study. A minimal set of screen failure information is required to ensure transparent reporting of screen failure participants to meet the Consolidated Standards of Reporting Trials (CONSORT) publishing requirements and to respond to queries from regulatory authorities. Minimal information includes demography, screen failure details, eligibility criteria, and any serious adverse event (SAE).

Individuals who do not meet the eligibility criteria for participation in this study may be considered for rescreening subject to sponsor's approval. Rescreened participants should be assigned a new participant number.



# 6. Study Intervention

Study intervention is defined as any investigational intervention(s), marketed product(s), placebo, or medical device(s) intended to be administered to a study participant according to the study protocol.

Study intervention will occur only on Day 1, and participants will not be retreated.

Participants will be observed at least 30 minutes after study intervention administration for AEs.

# 6.1. Study Intervention Administered



Approval Date: 12-Aug-2019

# CONFIDENTIAL

BOTOX





#### **BOTOX**

Table 6-2 Study Formulations and Dilution Instructions

| Study Intervention<br>Name | BOTOX High Dose | BOTOX Low Dose | Placebo |
|---|---|---|---|
| Packaging and<br>Labeling | Each study kit will have one vial powder. Each vial will be labeled as required. The high and low dose BOTOX | | Placebo vials will be supplied in kits with identical appearance to kits containing BOTOX vials. Each placebo vial will be labeled as required per country requirement. |
| Manufacturer | Allergan | | |

# 6.2. Preparation/Handling/Storage/Accountability

- 1. The investigator or designee must confirm appropriate temperature conditions have been maintained during transit for all study intervention received and any discrepancies are reported and resolved before use of the study intervention.
- 2. Only participants enrolled in the study may receive study intervention. Only the sponsor may supply the study intervention; only the Independent Drug Reconstitutor (IDR) may prepare the study intervention; and only the investigator, trained in the study-specific injection technique, may administer study intervention. All study intervention must be stored in a secure, environmentally controlled, and monitored (manual or automated) area in accordance with the labeled storage conditions with access limited to the investigator and authorized site staff.
- 3. The IDR is responsible for study intervention accountability, reconciliation, and record maintenance (ie, receipt, reconciliation, and final disposition records).
- 4. Further guidance and information for the final disposition of unused study interventions are provided in the Study Pharmacy Manual.



#### BOTOX

All unused study intervention and used kits must be returned to the sponsor at the termination of the study. Unit counts will be performed when the study intervention is returned, and all study intervention must be accounted for.

#### 6.3. Measures to Minimize Bias: Randomization and Blinding

At the Screening Visit (Visit 1), after the participant signs the ICF, the site will log on to the IWRS to obtain a participant number. At the time of randomization, eligible participants will be randomly assigned into 1 of the 3 treatment groups in a 1:1:1 allocation ratio to receive either BOTOX high dose, BOTOX low dose, or placebo, respectively (see Section 6.1). The automated IWRS will be used to manage the randomization and treatment assignment based on a randomization scheme prepared by the sponsor. The randomization will occur on Day 1 after all baseline procedures have been completed and the investigator has verified that the participant has met all inclusion and exclusion criteria.

At each study site, designated staff member(s) will serve as the IDR. This person will be unblinded and will be responsible for study intervention preparation and documentation. The IDR must not perform any other study-related procedures; and therefore, will have no role in participant evaluation, data entry, or in any efficacy or safety data collection, analyses, or assessment.

Study intervention will be labeled with kit numbers. The IWRS will provide the IDR with the specific kit number for each randomized participant at the time of randomization (Day 1). The IDR will dispense study intervention according to the IWRS. The IDR will receive the IWRS confirmation notifications for each transaction and will maintain these with the other unblinded study source documents with restricted access to the blinded site study staff. The IDR will prepare the study intervention as described in Table 6-2. Once the study intervention is reconstituted, the IDR will draw the required volume into an appropriately sized syringe and label the syringe with the participant's IWRS assigned ID number (and other information as specified in the Study Pharmacy Manual). All study intervention will be provided in identical syringes to maintain blinding of the study. The IDR will then provide the filled syringes to the investigator, who will inject the participant according to the study treatment administration instructions in Section 6.1.

Blinding is critical to the integrity of the clinical trial. The IWRS will be programmed with blind-breaking instructions. In case of an emergency, the investigator has the sole responsibility for determining if unblinding of a participant's study intervention assignment is warranted. Participant safety must always be the first consideration in making such a determination. If the investigator decides that unblinding is warranted, the investigator should make every effort to contact the sponsor prior to unblinding a participant's study intervention assignment unless this could delay emergency treatment of the participant. If a participant's study intervention



#### BOTOX

assignment is unblinded, the sponsor must be notified within 24 hours after breaking the blind. The date and reason that the blind was broken must be recorded in the source documentation.

#### **6.4.** Study Intervention Compliance

Participants will receive a single treatment of BOTOX under the direct supervision of study site personnel.

The study site will keep an accurate drug disposition record that specifies the amount of study intervention administered to each participant and the date of administration.

## 6.5. Concomitant Therapy

Study center staff must notify the sponsor immediately if a participant consumes any concomitant medications not permitted by the protocol. Participants who admit to using prohibited concomitant medications may be discontinued from the study at the discretion of the investigator or the sponsor.

The use of any concomitant medication or vaccine, (including prescription or over-the-counter medication, vitamins and/or herbal supplements), is to be recorded on the participant's eCRF at each visit along with the reason the medication is taken.

Concomitant therapy and/or medications considered necessary for the study participant's welfare may be given at the discretion of the investigator.

If concomitant medications may have an effect on efficacy or safety outcomes, these medications should be administered in dosages that remain constant throughout the course of the trial at the discretion of the investigator.

If the permissibility of a specific medication/treatment is in question, please contact the sponsor.

#### 6.5.1. Prohibited Interventions and Washout Before the Study

Refer to eligibility criteria (exclusion criteria, Section 5.2).

#### 6.5.2. Permitted Interventions

Any medication or vaccine (including over-the-counter or prescription medicines, vitamins, and/or herbal supplements) that the participant is receiving at the time of enrollment or receives during the study must be recorded along with:

- Indication/reason for medication use
- Dates of administration including start and end dates
- Dosage information including dose and frequency

Therapy considered necessary for the participant's welfare may be given at the discretion of the investigator. If the permissibility of a specific concomitant or prior medication/treatment is in question, please contact the sponsor.



#### BOTOX

Any medication taken during the study between the date of study intervention and the date of the EOS visit will be recorded in the eCRF as a concomitant medication; any medication started after the EOS visit will not be considered a concomitant medication and should not be captured in the eCRF.

#### 6.5.3. Prohibited Interventions During the Study

The decision to administer a prohibited medication/treatment during the study period is done with the safety of the study participant as the primary consideration. When possible, the sponsor is to be notified before the prohibited medication/treatment is administered.



#### 6.6. Dose Modification

No dose modifications are permitted.

# 6.7. Intervention after the End of the Study

No interventions after the end of study are planned.

# 7. Discontinuation of Study Intervention and Participant Discontinuation/Withdrawal

A premature discontinuation will occur if a participant who signs the ICF and is randomized ceases participation in the study, regardless of circumstances, before the completion of the protocol-defined study procedures.



#### **BOTOX**

Notification of early participant discontinuation from the study and the reason for discontinuation will be made to the sponsor and will be clearly documented in the appropriate eCRF.

The sponsor should be consulted in advance of withdrawal whenever possible. Every effort should be made to retain participants in the study until completion as much as possible. Participants who are withdrawn from the study may not be re-enrolled but will be asked to undergo all early withdrawal activities. Definitions of the standard terms are provided in Appendix 5.

Reasons for discontinuation from the study treatment and/or the study may include the following commonly used or other acceptable terms:

| Commonly Used Terms | Other Acceptable Terms |
|-----------------------------|------------------------|
| Adverse event | Death |
| Completed | |
| Lost to follow-up | |
| Other | |
| Physician decision | |
| Pregnancy | |
| Protocol deviation | |
| Screen failure | |
| Site terminated by sponsor | |
| Study terminated by sponsor | |
| Withdrawal by subject | |

# 7.1. Discontinuation of Study Intervention

If a participant does not tolerate study injections, the participant will be observed until the intolerability has either resolved or satisfactorily stabilized in the judgement of the investigator and the participant may choose to exit the study or to remain in the study for all safety follow-up assessments through the EOS Visit.

If a pregnancy is confirmed after the participant has received study intervention, the participant may choose to exit the study after appropriate safety follow-up or to remain in the study for all safety and efficacy follow-up assessments through the EOS visit.

# 7.2. Participant Discontinuation/Withdrawal from the Study

• A participant may withdraw from the study at any time at his/her own request or may be withdrawn at any time at the discretion of the investigator for safety, behavioral, compliance, or administrative reasons.



#### **BOTOX**

- If the participant withdraws consent for disclosure of future information, the sponsor may retain and continue to use any data collected before such a withdrawal of consent.
- See the SoA for data to be collected at the time of study discontinuation and follow-up and for any further evaluations that need to be completed.

## 7.3. Lost to Follow Up

A participant will be considered lost to follow-up if he/she repeatedly fails to return for scheduled visits and is unable to be contacted by the study site.

The following actions must be taken if a participant fails to return to the clinic for a required study visit:

- The site must attempt to contact the participant and reschedule the missed visit as soon as possible and counsel the participant on the importance of maintaining the assigned visit schedule and ascertain whether or not the participant wishes to and/or should continue in the study.
- Before a participant is deemed lost to follow-up, the investigator or designee must make every effort to regain contact with the participant (where possible, 3 telephone calls and, if necessary, a certified letter to the participant's last known mailing address or local equivalent methods). These contact attempts will be documented in the participant's medical record.
- Should the participant continue to be unreachable, he/she will be considered to have withdrawn from the study.

# 8. Study Assessments and Procedures

- Study procedures and their timing are summarized in the SoA (Section 1.2).
- Protocol waivers or exemptions are not allowed.
- Immediate safety concerns should be discussed with the sponsor immediately upon occurrence or awareness to determine if the participant should continue or discontinue study intervention.
- Adherence to the study design requirements, including those specified in the schedule of assessments, is essential and required for study conduct.
- All screening evaluations must be completed and reviewed to confirm that potential
  participants meet all eligibility criteria. The investigator will maintain a screening log to
  record details of all participants screened and to confirm eligibility or record reasons for
  screening failure, as applicable. During the Screening Period, the investigator or
  subinvestigator will assess the clinical significance of any physical examination findings.
  Any participants with abnormalities judged to meet exclusion criteria will be excluded from
  the study.



#### BOTOX

# 8.1. Efficacy Assessments

## 8.1.1. Primary Efficacy Assessment

Prior to enrolling participants, investigators (or subinvestigators when applicable) will be trained in grading platysma prominence severity using the C-APPS.



## 8.1.2. Secondary Efficacy Assessment





# CONFIDENTIAL Protocol 1936-201-008 Amd 1 BOTOX











# 8.2. Safety Assessments

Planned timepoints for all safety assessments are provided in the SoA (Section 1.2).



#### 8.2.2. Vital Signs

Vital signs will be assessed as follows:

Pulse rate, blood pressure, and respiratory rate will be assessed with participants in a sitting position; use of either a manual or automated device is acceptable.

- Pulse rate (beats per minute): Participants are to be seated for at least 5 minutes, and
  pulse will be counted over 60 seconds and recorded in the source document and eCRF as
  beats per minute.
- Blood pressure (mm Hg): Participants are to be seated for at least 5 minutes and systolic and diastolic blood pressure will be measured.
- Respiration rate (breaths per minute): Participants are to be seated for at least 5 minutes and breaths will be counted for 30 seconds and multiplied by 2.

#### 8.2.3. Pregnancy Testing

Women of childbearing potential (WOCBP) must have a negative urine test result before receiving study intervention. A urine pregnancy test may also be performed at any other visit, at the investigator's discretion.

#### 8.3. Adverse Events and Serious Adverse Events

The definitions of an AE or SAE can be found in Appendix 3.

AEs will be reported by the participant (or, when appropriate, by a caregiver or surrogate).


#### **BOTOX**

The investigator and any qualified designees are responsible for collecting, detecting, documenting, and recording events that meet the definition of an AE or SAE and any other study-specific term as relevant and remain responsible for following up AEs that are serious, considered related to the study intervention or study procedures, or that caused the participant to discontinue the study (see Section 7).

## 8.3.1. Time Period and Frequency for Collecting Adverse Event and Serious Adverse Event Information

All SAEs from the signing of the ICF until the follow-up visit will be collected at the timepoints specified in the SoA (Section 1.2), and as observed or reported spontaneously by study participants.

All AEs from the signing of the ICF until the follow-up visit will be collected at the timepoints specified in the SoA (Section 1.2), and as observed or reported spontaneously by study participants.

Medical occurrences that begin before the start of study intervention, but after obtaining informed consent will be recorded in the AE section of the eCRF.

All SAEs will be recorded and reported to the sponsor or designee within 24 hours of awareness, as indicated in Appendix 3. The investigator will submit any updated SAE data to the sponsor within 24 hours of it being available.

AESIs are described below in Section 8.3.6 and in Appendix 3.

Investigators are not obligated to actively seek AE or SAE information after conclusion of the study participation. However, if the investigator learns of any SAE, including a death, at any time after a participant has been discharged from the study, and he/she considers the event to be reasonably related to the study intervention or study participation, the investigator must promptly notify the sponsor.

The method of recording, evaluating, and assessing causality of AEs and SAEs and the procedures for completing and transmitting SAE reports are provided in Appendix 3.

#### 8.3.2. Method of Detecting Adverse Events and Serious Adverse Events

Care will be taken not to introduce bias when detecting AEs and/or SAEs. Open-ended and non-leading verbal questioning of the participant is the preferred method to inquire about AE occurrences.

#### 8.3.3. Follow-up of Adverse Events and Serious Adverse Events

After the initial AE/SAE report, the investigator is required to proactively follow each participant at subsequent visits/contacts. All SAEs and AESI (as defined in Section 8.3.6) will be followed until resolution, stabilization, the event is otherwise explained, or the participant is lost to follow-up (as defined in Section 7.3).



#### **BOTOX**

The investigator is obligated to perform or arrange for the conduct of supplemental measurements and/or evaluations as medically indicated or as requested by the sponsor to elucidate the nature and/or causality of the AE or SAE as fully as possible. This may include additional laboratory tests or investigations, histopathological examinations, or consultation with other health care professionals.

If a participant dies during participation in the study or during a recognized follow-up period, the investigator will provide the sponsor with a copy of any postmortem findings including histopathology.

New or updated information will be recorded in the originally completed eCRF.

The investigator will submit any updated SAE data to the sponsor within 24 hours of receipt of the information.

#### 8.3.4. Regulatory Reporting Requirements for Serious Adverse Events

- Prompt notification by the investigator to the sponsor of an SAE is essential so that legal obligations and ethical responsibilities towards the safety of participants and the safety of a study intervention under clinical investigation are met.
- The sponsor has a legal responsibility to notify both the local regulatory authority and other regulatory agencies about the safety of a study intervention under clinical investigation. The sponsor will comply with country-specific regulatory requirements relating to safety reporting to the regulatory authority, IRBs/ IECs, and investigators.
- Investigator safety reports must be prepared for SUSARs according to local regulatory requirements and sponsor policy and forwarded to investigators as necessary.
- An investigator who receives an investigator safety report describing an SAE or other specific safety information (eg, summary or listing of SAEs) from the sponsor will review and then file it along with the IB and will notify the IRB/IEC, if appropriate according to local requirements.

#### 8.3.5. Pregnancy

- Details of all pregnancies in female participants will be collected after the start of study intervention and until the EOS.
- If a pregnancy is reported, the investigator should inform the sponsor within 24 hours of learning of the pregnancy and should follow the procedures outlined in Appendix 7.
- Abnormal pregnancy outcomes (eg, spontaneous or elective abortion, fetal death, stillbirth, congenital anomalies, ectopic pregnancy) are considered SAEs.





#### 8.3.7. Medication Errors

Medication error refers to any unintended error in the dosing and/or administration of the study intervention as per instructions in the protocol, for example:

- Wrong study intervention
- Wrong dose (including dosing regimen, strength, form, concentration, amount)
- Wrong route of administration
- Wrong participant (ie, not administered to the intended participant)

#### **8.4.** Treatment of Overdose

The LD<sub>50</sub> for BOTOX in humans is estimated from primate studies to be approximately 3000 U. This makes accidental injection of a lethal dose highly unlikely, but significant AEs may still occur at doses below the LD<sub>50</sub> (Herrero 1967, Scott 1989).

Excessive doses may produce local or distant, generalized, and profound neuromuscular paralysis. Should accidental injection or oral ingestion occur or overdose be suspected, the participant should be medically monitored for up to several weeks for progressive signs or symptoms of systemic muscular weakness that could be local or distant from the site of injection, and which may include ptosis, diplopia, dysphagia, dysarthria, generalized weakness, or respiratory failure.

If the musculature of the oropharynx and esophagus is affected, aspiration may occur, which may lead to development of aspiration pneumonia. If the respiratory muscles become paralyzed or sufficiently weakened, intubation and assisted respiration may be necessary until recovery takes place. Supportive care could involve the need for a tracheostomy and/or prolonged mechanical ventilation, in addition to other general supportive care. Additional information is available in the IB.

Approval Date: 12-Aug-2019





#### BOTOX

In the event of an overdose, the investigator should:

- 1. Contact the sponsor immediately.
- 2. Closely monitor the participant for any AE/SAE and seek medical help as needed.
- 3. Document the quantity of the excess dose as well as the duration of the overdose in the eCRF as well as other details that led to the overdose.

#### 8.5. Pharmacokinetics

Pharmacokinetic parameters are not evaluated in this study.

#### 8.6. Pharmacodynamics

Pharmacodynamic parameters are not evaluated in this study.

#### 8.7. Genetics

Genetics are not evaluated in this study.

#### 8.8. Biomarkers and Other Assessments

Biomarkers are not evaluated in this study.

#### 8.9. Health Economics

Health economics are not evaluated in this study.







## 9.2. Sample Size Determination



Approximately 165 participants will be enrolled in a 1:1:1 randomization allocation ratio, yielding approximately 55 participants in the BOTOX high dose group, 55 participants in the BOTOX low dose group, and 55 participants in the placebo group.



## 9.3. Populations for Analyses

The 2 analysis populations are defined below:

 The mITT population includes all randomized participants with ≥ 1 postbaseline assessment for the primary efficacy endpoint. Participants will be summarized according to the randomized study intervention.



#### **BOTOX**

 The safety population includes all randomized participants who are administered study intervention. Participants will be summarized according to the study intervention they received.

#### 9.4. Statistical Analyses

The SAP and PRO SAP for psychometric analysis will be developed and finalized before database lock and will describe the participant populations to be included in the analyses, and procedures for accounting for missing, unused, and spurious data. This section summarizes the main features of the planned statistical analyses of the primary and secondary endpoints.

#### 9.4.1. Efficacy Analyses

#### 9.4.1.1. Primary and Secondary Endpoints

The primary and secondary efficacy endpoints will be analyzed for the mITT population (Table 9-2). All other efficacy endpoints and analyses will be defined in the SAP.

Table 9-2 Primary and Secondary Endpoints

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| C-APPS Responder (primary endpoint) | Achievement of ≥ 1-grade C-APPS improvement at maximum contraction at Day 14 | Day 14 | Responder |
| P-APPS Responder (secondary endpoint) | Achievement of ≥ 1-grade P-APPS improvement at maximum contraction at Day 14 | Day 14 | Responder |

#### 9.4.1.2. Multiple Comparisons Procedure

The overall FWER will be controlled at  $\alpha = 0.05$  for the set of primary and secondary endpoint comparisons between each of the BOTOX groups versus placebo (4 comparisons). The overall serial gatekeeping MCP will be used to control FWER and is defined in Table 9-3.

Table 9-3 Multiple Comparisons Procedure

| MCP Step <sup>a</sup> | Endpoint | MCP Criteria |
|---|---|---|
| 1 | C-APPS responder (BOTOX high dose vs placebo) | Nominal p-value $\leq \alpha$ |
| 2 | P-APPS responder (BOTOX high dose vs placebo) | Nominal p-value $\leq \alpha$ |
| 3 | C-APPS responder (BOTOX low dose vs placebo) | Nominal p-value $\leq \alpha$ |
| 4 | P-APPS responder (BOTOX low dose vs placebo) | Nominal p-value $\leq \alpha$ |

<sup>&</sup>lt;sup>a</sup> Serial gatekeeping MCP only proceeds to next step if all endpoints are statistically significant after application of MCP criteria in previous and current MCP steps for a BOTOX group.



**BOTOX** 

#### 9.4.1.3. Primary and Secondary Analyses

The proportion of responders will be analyzed using CMH tests.

In addition, 2-sided 95% confidence intervals for the treatment differences in response rates will be provided. Between group comparisons will only be performed for each BOTOX group against the placebo group, and BOTOX high dose group against the BOTOX low dose group.

#### 9.4.2. Safety Analyses

The safety analyses will be performed using the safety population and will be fully defined in the SAP. The safety parameters will include AEs and vital signs. For each safety parameter, the last nonmissing safety assessment before the first dose of study intervention will be used as the baseline for all analyses of that safety parameter.

#### 9.4.2.1. Adverse Events

An AE will be considered a TEAE if:

- The AE began after the first dose of study intervention; or
- The AE was present before the first dose of study intervention, but increased in severity or became serious after the first dose of study intervention

An AE will be considered a serious TEAE if it is a TEAE that additionally meets any SAE criteria.

The total number and percentage of participants reporting AEs, TEAEs, treatment-related TEAEs, serious TEAEs, treatment-related serious TEAEs, deaths, and discontinuations due to TEAEs will be summarized for each treatment group.

The number and percentage of participants reporting TEAEs in each study intervention group will be tabulated by system organ class, preferred term, and severity.

The number and percentage of participants reporting serious TEAEs in each study intervention group will be tabulated by system organ class and preferred term.

The number and percentage of participants reporting treatment-related TEAEs in each study intervention group will be tabulated by system organ class and preferred term.

If more than 1 AE is coded to the same PT for the same participant, the participant will be counted only once for that preferred term using the most severe and most related occurrence for the summarizations by severity and by relationship to study intervention.

The number and percentage of participants reporting TEAEs that are included in the possible distant spread of toxin (PDSOT) term list in each study intervention group will be tabulated by preferred term. The PDSOT term list will be provided by the medical safety physician (MSP).

The PDSOT will be reviewed by the MSP on a monthly basis for monitoring severity, frequency, and trending.



#### BOTOX

Listings of all AEs, SAEs, and AEs leading to discontinuation by participant will be presented. The definitions of an AE and SAE can be found in Appendix 3.



#### 9.4.2.3. Vital Signs

Descriptive statistics for vital signs (systolic and diastolic BP, pulse rate, and respiration rate) at baseline and changes from baseline at each assessment will be presented by study intervention.

#### 9.4.3. Other Analyses

All other exploratory efficacy analyses will be described in the SAP. Psychometric analysis will be performed by a CRO and described in a separate PRO SAP.

#### 9.5. Interim Analyses

Interim analyses are not planned for this study.



#### 10. Supporting Documentation and Operational Considerations

## 10.1. Appendix 1: Regulatory, Ethical, and Study Oversight Considerations

#### 10.1.1. Regulatory and Ethical Considerations

- This study will be conducted in accordance with the protocol and with the following:
  - Consensus ethical principles derived from international guidelines including the Declaration of Helsinki and CIOMS International Ethical Guidelines
  - o Applicable ICH/ISO/GCP guidelines
  - o Applicable laws and regulations
- The protocol, protocol amendments, ICF, IB, and other relevant documents (eg, advertisements) must be submitted to an IRB/IEC by the investigator and reviewed and approved by the IRB/IEC before the study is initiated.
- Any amendments to the protocol will require IRB/IEC approval before implementation of changes made to the study design, except for changes necessary to eliminate an immediate hazard to study participants.
- The investigator will be responsible for the following:
  - Providing written summaries of the status of the study to the IRB/IEC annually or more frequently in accordance with the requirements, policies, and procedures established by the IRB/IEC
  - Notifying the IRB/IEC of SAEs or other significant safety findings as required by IRB/IEC procedures
  - Providing oversight of the overall conduct of the study at the site and adherence to requirements of applicable local regulations, for example 21 CFR, ICH guidelines, the IRB/IEC, and European regulation 536/2014 for clinical studies (if applicable)

#### 10.1.2. Financial Disclosure

Investigators and subinvestigators will provide the sponsor with sufficient, accurate financial information as requested to allow the sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate regulatory authorities. Investigators are responsible for providing information on financial interests during the study and for 1 year after completion of the study.



#### **BOTOX**

#### 10.1.3. Informed Consent Process

- The investigator or his/her representative will explain the nature of the study to the participant and answer all questions regarding the study.
- Participants must be informed that their participation is voluntary. Participants will be
  required to sign a statement of informed consent that meets the requirements of 21 CFR 50,
  local regulations, ICH guidelines, HIPAA requirements, where applicable, and the IRB/IEC
  or study center.
- The medical record must include a statement that written informed consent was obtained before the participant was enrolled in the study and the date the written consent was obtained. The authorized person obtaining the informed consent must also sign the ICF.
- Participants must be re-consented to the most current version of the ICF(s) during their participation in the study.
- A copy of the ICF(s) must be provided to the participant or the participant's legally authorized representative.
- Participants who are rescreened are not required to sign a new ICF if rescreening occurs within 14 days of first signing the ICF.

#### 10.1.4. Data Protection

- Participants will be assigned a unique identifier. Any participant records, datasets, or photographs that are transferred to the sponsor will contain the identifier only; participant names or any information which would make the participant identifiable will not be transferred.
- The participant must be informed that his/her personal study-related data will be used by the sponsor in accordance with local data protection law. The level of disclosure must also be explained to the participant.
- The participant must be informed that his/her medical records may be examined by Clinical Quality Assurance auditors or other authorized personnel appointed by the sponsor, by appropriate IRB/IEC members, and by inspectors from regulatory authorities.

#### 10.1.5. Posting Clinical Study Data

- Company-sponsored study information and tabular study results will be posted to the US National Institutes of Health website www.clinicaltrials.gov and other publicly accessible sites, if applicable.
- Study data and information may be published in non-promotional, peer-reviewed publications either by or on behalf of the sponsor.
- Clinical study reports, safety updates and annual reports will be provided to regulatory authorities as required.



#### **BOTOX**

#### 10.1.6. Data Quality Assurance

- All participant data relating to the study will be recorded on printed or eCRFs unless transmitted to the sponsor or designee electronically. The investigator is responsible for verifying that data entries are accurate and correct by electronically signing the eCRF.
- The investigator must maintain accurate documentation (source data) that supports the information entered in the eCRF.
- The investigator must permit study-related monitoring, audits, IRB/IEC review, and regulatory agency inspections and provide direct access to source data documents.
- The sponsor or designee is responsible for the data management of this study including quality checking of the data.
- Study monitors will perform ongoing source data verification to confirm that data entered into the CRF by authorized site personnel are accurate, complete, and verifiable from source documents; that the safety and rights of participants are being protected; and that the study is being conducted in accordance with the currently approved protocol and any other study agreements, ICH GCP, and all applicable regulatory requirements.
- Records and documents, including signed ICFs, pertaining to the conduct of this study must be retained by the investigator as stated in the clinical trial agreement. No records may be destroyed during the retention period without the written approval of the sponsor. No records may be transferred to another location or party without written notification to the sponsor.

#### **10.1.7.** Source Documents

- Source documents provide evidence for the existence of the participant and substantiate the integrity of the data collected. Source documents are filed at the investigator's site.
- Data entered in the eCRF that are transcribed from source documents must be consistent with the source documents or the discrepancies must be explained. The investigator may need to request previous medical records or transfer records, depending on the study. Also, current medical records must be available.
- Definition of what constitutes source data can be found in Section 4.0 of ICH E6, Good Clinical Practice: Consolidated Guidance and must follow ALCOA, ie, records must be attributable, legible, contemporaneous, original, and accurate.
- Source data are defined as: original documents, data, and records (eg, hospital records, clinical and office charts, diaries or evaluation checklists, pharmacy dispensing records, recorded data from automated instruments, copies or transcriptions certified after verification as being accurate and complete, microfiche, photographic images, negatives, microfilm or magnetic media, X-rays, participant files, and records kept at the pharmacy, at the laboratories, and at medico-technical departments involved in the clinical study). These records include, but are not limited to, original signed and dated consent forms, relevant



#### **BOTOX**

observations including records of AEs, and records of all exposure to study intervention, and data entered directly into an eCOA device.

- The following information should be entered into the participant's source records, including but not limited to:
  - O Statement that standardized photographs were taken as appropriate and data images submitted to the designated third-party vendor
  - Pregnancy test results for WOCBP

#### 10.1.8. Study and Site Closure

The sponsor designee reserves the right to close the study site or terminate the study at any time for any reason at the sole discretion of the sponsor. Study sites will be closed upon study completion. A study site is considered closed when all required documents and study supplies have been collected and a study-site closure visit has been performed.

The investigator may initiate study-site closure at any time, provided there is reasonable cause and sufficient notice is given in advance of the intended termination.

Reasons for the early closure of a study site by the sponsor or investigator may include but are not limited to:

- Failure of the investigator to comply with the protocol, the requirements of the IRB/IEC or local health authorities, the sponsor's procedures, or GCP guidelines
- Inadequate recruitment of participants by the investigator
- Discontinuation of further development of study intervention

#### 10.1.9. Publication Policy

- Allergan as the sponsor has proprietary interest in this study. Authorship and manuscript composition will reflect joint cooperation between multiple investigators and sites and Allergan personnel. Authorship will be established prior to the writing of the manuscript. As this study involves multiple centers, no individual publications will be allowed prior to completion of the final report of the multicenter study except as agreed with Allergan.
- The sponsor will comply with the requirements for publication of study results. In accordance with standard editorial and ethical practice, the sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data.
- Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

#### 10.1.10. Compliance with Protocol

The investigator is responsible for compliance with the protocol at the investigational site. A representative of the sponsor will make frequent contact with the investigator and his/her research staff and will conduct regular monitoring visits at the site to review participant and



Protocol 1936-201-008 Amd 1

#### **BOTOX**

study intervention accountability records for compliance with the protocol. Protocol deviations will be discussed with the investigator upon identification. The use of the data collected for the participant will be discussed to determine if the data are to be included in the analysis. The investigator will enter data that may be excluded from analysis as defined by the protocol deviation specifications. Significant protocol deviations will be reported to the IRB/IEC according to the IRB/IEC's reporting requirements.



# **10.2. Appendix 2: Clinical Laboratory Tests** Not applicable.



## 10.3. Appendix 3: Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting

#### **Definition of AE**

#### **AE Definition**

- An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
- An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention.

#### AE of Special Interest (AESI)

An AESI is an AE of scientific and medical concern specific to the sponsor's study drug/device or program, which warrants ongoing monitoring and rapid communication by the investigator to the sponsor. Such an event might warrant further investigation in order to characterize and understand it.

Dysphagia, dyspnea, aspiration, and aspiration pneumonia have been identified as AESIs for the study intervention in this protocol.

Upon identification and awareness of 1 or more of these events, the investigator must document and report the event by completing an AE eCRF, and must notify the MSP and assigned Regional Site Manager by email or phone call within 72 hours of awareness. The SAE/AESI form is not needed unless the AESI is serious.

If the AESI meets SAE criteria (which are listed below), it will be reported within 24 hours of awareness per the sponsor's SAE reporting requirements (described below).

#### **Events Meeting the AE Definition**

- Any safety assessments (eg, vital signs measurements), including those that worsen from baseline, considered clinically significant in the medical and scientific judgment of the investigator (ie, not related to progression of underlying disease). The test result is considered to be an AE by the investigator or sponsor.
- Exacerbation of a chronic or intermittent pre-existing condition including either an increase in frequency and/or intensity of the condition
- New condition detected or diagnosed after study intervention administration even though it may have been present before the start of the study
- Signs, symptoms, or the clinical sequelae of a suspected drug-drug interaction



#### BOTOX

- Signs, symptoms, or the clinical sequelae of a suspected overdose of either study intervention or a concomitant medication. Overdose per se will not be reported as an AE or SAE unless it is an intentional overdose taken with possible suicidal/self-harming intent. Such overdoses should be reported regardless of sequelae.
- Lack of efficacy or failure of expected pharmacological action per se will not be reported
  as an AE or SAE. Such instances will be captured in the efficacy assessments. However,
  the signs, symptoms, and/or clinical sequelae resulting from lack of efficacy will be
  reported as AEs or SAEs if they fulfil the definition of an AE or SAE.

#### Events NOT Meeting the AE Definition

- Any clinically significant abnormal laboratory findings or other abnormal safety
  assessments that are associated with the underlying disease, unless judged by the
  investigator to be more severe than expected for the participant's condition. Merely
  repeating an abnormal test, in the absence of any of the above conditions, does not
  constitute an AE. Any abnormal test result that is determined to be an error does not
  require recording as an AE.
- The disease/disorder being studied or expected progression, signs, or symptoms (clearly defined) of the disease/disorder being studied, unless more severe than expected for the participant's condition
- Medical or surgical procedure (eg, endoscopy, appendectomy): the condition that leads to the procedure is the AE
- Situations in which an untoward medical occurrence did not occur (social and/or convenience admission to a hospital)
- Anticipated day-to-day fluctuations of pre-existing disease(s) or condition(s) present or detected at the start of the study that do not worsen



#### **BOTOX**

#### **Definition of SAE**

SAEs must meet both the AE criteria described above and the seriousness criteria listed below.

#### An SAE is defined as any untoward medical occurrence that, at any dose:

#### a. Results in death

#### b. Is life threatening

The term *life threatening* in the definition of *serious* refers to an event in which the participant was at risk of death at the time of the event. It does not refer to an event, which hypothetically might have caused death, if it were more severe.

#### c. Requires inpatient hospitalization or prolongation of existing hospitalization

In general, hospitalization signifies that the participant has been detained (usually involving at least an overnight stay) at the hospital or emergency ward for observation and/or intervention that would not have been appropriate in the physician's office or outpatient setting. Complications that occur during hospitalization are AEs. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether hospitalization occurred or was necessary, the AE should be considered serious.

Hospitalization for elective intervention of a pre-existing condition that did not worsen from baseline is not considered an AE.

#### d. Results in persistent disability/incapacity

- The term disability means a substantial disruption of a person's ability to conduct normal life functions.
- This definition is not intended to include experiences of relatively minor medical significance such as uncomplicated headache, nausea, vomiting, diarrhea, influenza, and accidental trauma (eg, sprained ankle) which may interfere with or prevent everyday life functions but do not constitute a substantial disruption.

#### e. Is a congenital anomaly/birth defect

#### f. Other situations:

 Medical or scientific judgment should be exercised in deciding whether SAE reporting is appropriate in other situations such as important medical events that may not be immediately life threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition. These events should usually be considered serious.

Examples of such events include invasive or malignant cancers, intensive intervention in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization, or development of drug dependency or drug abuse.



BOTOX

### Recording and Follow-Up of AEs and/or SAEs

#### AE and SAE Recording

- When an AE or SAE occurs, it is the responsibility of the investigator to review all
  documentation (eg, hospital progress notes, laboratory reports, and diagnostics reports)
  related to the event.
- The investigator will then record all relevant AE or SAE information in the eCRF.
- It is **not** acceptable for the investigator to send photocopies of the participant's medical records to the sponsor in lieu of completion of the AE or SAE eCRF page.
- There may be instances when copies of medical records for certain cases are requested by the sponsor. In this case, all participant identifiers, with the exception of the participant number, will be redacted on the copies of the medical records before submission to the sponsor.
- The investigator will attempt to establish a diagnosis of the event based on signs, symptoms, and/or other clinical information. Whenever possible, the diagnosis (not the individual signs/symptoms) will be documented as the AE/SAE.

## Assessment of Intensity

| MILD | A type of AE that is usually transient and may require only minimal treatment or therapeutic intervention. The event does not generally interfere with usual activities of daily living. |
|---|---|
| MODERATE | A type of AE that is usually alleviated with additional specific therapeutic intervention. The event interferes with usual activities of daily living, causing discomfort but poses no significant or permanent risk of harm to the research participant. |
| SEVERE | A type of AE that interrupts usual activities of daily living, or significantly affects clinical status, or may require intensive therapeutic intervention. |

An event is defined as *serious* when it meets at least one of the predefined outcomes as described in the definition of an SAE, NOT when it is rated as severe.



#### BOTOX

#### **Assessment of Causality**

- The investigator is obligated to assess the relationship between study intervention and each occurrence of each AE or SAE.
- A reasonable possibility of a relationship conveys that there are facts, evidence, and/or
  arguments to suggest a causal relationship, rather than a relationship cannot be ruled out.
- The investigator will use clinical judgment to determine the relationship.
- Alternative causes, such as underlying disease(s), concomitant therapy, and other risk factors, as well as the temporal relationship of the event to study intervention administration will be considered and investigated.
- The investigator will also consult the IB and/or product information, for marketed products, in his/her assessment.
- For each AE or SAE, the investigator <u>must</u> document in the medical notes that he/she has reviewed the AE or SAE and has provided an assessment of causality.
- There may be situations in which an SAE has occurred and the investigator has minimal information to include in the initial report to the sponsor. However, it is very important that the investigator always make an assessment of causality for every event before the initial transmission of the SAE data to the sponsor.
- The investigator may change his/her opinion of causality in light of follow-up information and send an SAE follow-up report with the updated causality assessment.
- The causality assessment is one of the criteria used when determining regulatory reporting requirements.

#### Reporting of SAEs

#### **SAE Reporting**

- Email is the preferred method to transmit SAE information. The email address is IR-Clinical-SAE@allergan.com.
- Facsimile transmission of the SAE information is also acceptable. The fax number is +1-714-796-9504 (backup number is +1-714-246-5295).
- In rare circumstances and in the absence of facsimile equipment, notification by telephone is acceptable with a copy of the SAE form, sent by overnight mail or courier service.
- Initial notification via telephone does not replace the need for the investigator to complete and sign the SAE form within the designated reporting time frames.
- Contacts for SAE reporting can be found on the protocol title page.



## 10.4. Appendix 4: Abbreviations

3D 3-dimensional

AE adverse event

ALCOA attributable, legible, contemporaneous, original, and accurate

BOTOX botulinum toxin type A purified neurotoxin

BP blood pressure

C-APPS Clinician Allergan Platysma Prominence Scale

CDISC Clinical Data Interchange Standards Consortium

CFR code of federal regulations

CIOMS Council for International Organizations of Medical Sciences

CMH Cochran-Mantel-Haenszel

CONSORT Consolidated Standards of Reporting Trials

CRO contract research organization

eCOA electronic clinical outcomes assessment (via tablet)

eCRF electronic case report form

EDC electronic data capture

EOS end of study

FWER familywise error rate GCP good clinical practice

HEENT head, eyes, ears, nose, throat

HIPAA Health Insurance Portability and Accountability Act of 1996

IB investigator's brochure ICF informed consent form

ICH International Council on Harmonisation

IDR independent drug reconstitutor
IEC independent ethics committee

IND Investigational New Drug



Protocol 1936-201-008 Amd 1

**BOTOX** 

IRB institutional review board

ISO International Organization for Standardization

IWRS Interactive Web Response System

MCP multiple comparisons procedure

mITT modified intent-to-treat

MSP medical safety physician

NCI National Cancer Institute

P-APPS Participant Allergan Platysma Prominence Scale

PDSOT possible distant spread of toxin

PRO patient reported outcome

PT preferred term

SAE serious adverse event
SAP statistical analysis plan
SoA Schedule of Activities

SUSAR suspected unexpected serious adverse reactions

TEAE treatment-emergent adverse event WOCBP woman of childbearing potential



## 10.5. Appendix 5: Standard Discontinuation Criteria

This table provides participant discontinuation criteria for this protocol. CDISC terminology is used, and thus *subject* or *patient* is used instead of *participant* (as used elsewhere in this protocol). These terms are interchangeable.

| CDISC Submission Value | CDISC Definition |
|---|---|
| Adverse event | Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. For further information, see the ICH Guideline for Clinical Safety Data Management: Definitions and Standards for Expedited Reporting (modified from ICH E2A) Synonyms: side effect, adverse experience. See also serious adverse event, serious adverse experience. (CDISC glossary) |
| Completed | To possess every necessary or normal part or component or step; having come or been brought to a conclusion (NCI) |
| Death | The absence of life or state of being dead (NCI) |
| Lost to follow-up | The loss or lack of continuation of a subject to follow-up |
| Other | Different than the one(s) previously specified or mentioned (NCI) |
| Physician decision | A position, opinion or judgment reached after consideration by a physician with reference to subject (NCI) |
| Pregnancy | Pregnancy is the state or condition of having a developing embryo or fetus in the body (uterus), after union of an ovum and spermatozoon, during the period from conception to birth. (NCI) |
| Protocol deviation | An event or decision that stands in contrast to the guidelines set out by the protocol (NCI) |
| Screen failure | The potential subject who does not meet one or more criteria required for participation in a trial |
| Site terminated by sponsor | An indication that a clinical study was stopped at a particular site by its sponsor (NCI) |
| Study terminated by sponsor | An indication that a clinical study was stopped by its sponsor (NCI) |
| Withdrawal by subject | An indication that a study participant has removed itself from the study (NCI) |



## 10.6. Appendix 6: Study Tabular Summary

This table is intended for use in posting study information to registries (eg, ClinicalTrials.gov).

| Parameter Group | Parameter | Value |
|---|---|---|
| Trial information | Trial Title | A Phase 2 Multicenter, Randomized,<br>Double-Blind, Placebo-Controlled, Dose-<br>Ranging Study to Evaluate the Safety and<br>Efficacy of BOTOX® (Botulinum Toxin<br>Type A) Purified Neurotoxin Complex for<br>the Treatment of Platysma Prominence |
| | Clinical Study Sponsor | Allergan Sales LLC |
| | Trial Phase Classification | Phase 2 |
| | Trial Indication | Platysma Prominence |
| | Trial Indication Type | Treatment |
| | Trial Type | Efficacy |
| | | Safety |
| | Trial Length | Approximately 4 months |
| | Planned Country of Investigational Sites | United States and Canada |
| | Planned Number of Subjects | 165 |
| | FDA-Regulated Device Study | No |
| | FDA-Regulated Drug Study | Yes |
| | Pediatric Study | No |
| Subject information | Diagnosis Group | Adults with moderate to severe platysma prominence |
| | Healthy Subject Indicator | Yes |
| | Planned Minimum Age of Subjects | 18 |
| | Planned Maximum Age of Subjects | No upper age limit |
| | Sex of Participants | Male or Female |
| | Stable Disease Minimum Duration | Not applicable |



| Parameter Group | Parameter | Value |
|---|---|---|
| Treatments | Investigational Therapy or Treatment | OnabotulinumtoxinA |
| | Intervention Type | Drug |
| | Pharmacological Class of Invest. Therapy | Neurotoxin |
| | Dose per Administration | Up to U |
| | Dose Units | U |
| | Dosing Frequency | Single-treatment on Day 1 |
| | Route of Administration | Intramuscular |
| | Current Therapy or Treatment | Not applicable |
| | Added on to Existing Treatments | No |
| | Control Type | Placebo |
| | Comparative Treatment Name | Not applicable |
| Trial design | Study Type | Interventional |
| | Intervention Model | Parallel |
| | Planned Number of Arms | 3 |
| | Trial is Randomized | Yes |
| | Randomization Quotient | 1:1:1 (BOTOX high dose:BOTOX low dose:placebo) |
| | Trial Blinding Schema | Double blind |
| | Adaptive Design | No |
| | Study Stop Rules | Not applicable |



## 10.7. Appendix 7: Contraceptive Guidance and Collection of Pregnancy Information

#### **Definitions:**

#### Woman of Childbearing Potential (WOCBP)

A woman is considered fertile following menarche and until becoming postmenopausal unless permanently sterile (see below).

#### Women in the following categories are not considered WOCBP:

- 1. Premenarchal
- 2. Premenopausal female with 1 of the following:
  - Documented hysterectomy
  - Documented bilateral salpingectomy
  - Documented bilateral oophorectomy

Note: Documentation can come from the site personnel's: review of the participant's medical records, medical examination, or medical history interview.

#### 3. Postmenopausal female

• A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle-stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy (HRT). However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.

#### **Contraception Guidance:**

#### **Female Participants**

Female participants of childbearing potential are eligible to participate if they agree to use a highly effective method or acceptable method of contraception consistently and correctly as described in Table 10–1.



#### **BOTOX**

#### Table 10-1 Highly Effective and Acceptable Contraceptive Methods

#### Highly Effective Contraceptive Methods That Are User Dependent<sup>a</sup>

Failure rate of < 1% per year when used consistently and correctly

Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation<sup>b</sup>

- Oral
- Intravaginal
- Transdermal

Progestogen-only hormonal contraception associated with inhibition of ovulation

- Oral
- Injectable

#### Highly Effective Methods That Are User Independent<sup>a</sup>

Implantable progestogen-only hormonal contraception associated with inhibition of ovulation

- Intrauterine device (IUD)
- Intrauterine hormone-releasing system (IUS)
- Etonogestrel implant (ie, Nexplanon®)

Bilateral tubal occlusion

Intrauterine copper contraceptive (ie, ParaGard®)

#### Vasectomized Partner

A vasectomized partner is a highly effective contraception method provided that the partner is the sole male sexual partner of the WOCBP and the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used.

#### Sexual Abstinence

Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study intervention. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant.

#### **Acceptable Methods**

Acceptable birth control methods that result in a failure of more than 1% per year include:

- Progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mode of action
- Male or female condom with or without spermicide
- Cap, diaphragm, or sponge with spermicide
- Nonhormonal intrauterine device

A combination of male condom with either cap, diaphragm, or sponge with spermicide (double-barrier methods) are also considered acceptable, but not highly effective, birth control methods.

<sup>a</sup> Typical use failure rates may differ from those when used consistently and correctly. Use should be consistent with local regulations regarding the use of contraceptive methods for participants participating in clinical studies.



**BOTOX** 

#### **Pregnancy Testing:**

- WOCBP should only be included after a confirmed menstrual period and a negative highly sensitive pregnancy test at screening and also a negative test on Day 1.
- Additional pregnancy testing may also be performed at any other study visit at the investigator's discretion and at the study exit visit, and as required locally.
- Pregnancy testing will be performed whenever a menstrual cycle is missed or when pregnancy is otherwise suspected.

#### **Collection of Pregnancy Information:**

#### Female Participants Who Become Pregnant

- The investigator will collect pregnancy information on any female participant who becomes pregnant while participating in this study. Information will be recorded on the appropriate form and submitted to the sponsor within 24 hours of learning of a participant's pregnancy. The participant will be followed to determine the outcome of the pregnancy. The investigator will collect follow-up information on the participant and the neonate, and the information will be forwarded to the sponsor. Generally, follow-up will not be required for longer than 6 to 8 weeks beyond the estimated delivery date. Any termination of pregnancy will be reported, regardless of fetal status (presence or absence of anomalies) or indication for the procedure.
- While pregnancy itself is not considered to be an AE or SAE, any pregnancy complication will be reported as an AE or SAE. A spontaneous or elective abortion is always considered to be an SAE and will be reported as such. Any poststudy pregnancy-related SAE considered reasonably related to the study intervention by the investigator will be reported to the sponsor as described in Section 8.3.4. While the investigator is not obligated to actively seek this information in former study participants, he or she may learn of an SAE through spontaneous reporting.
- If a pregnancy is confirmed after the participant has received study intervention, the participant may choose to exit the study after appropriate safety follow-up or to remain in the study for all safety and efficacy follow-up assessments through the end-of-study visit.



## 10.8. Appendix 8: Clinician Allergan Platysma Prominence Scale

C-APPS grades and descriptions are shown in Section 8.1.1, Table 8-1.



10.9.









## 10.10. Appendix 10: Example Patient-Reported Outcomes Questionnaires, Descriptions, and Instructions

This appendix provides complete samples of each questionnaire; however, participants will provide responses in electronic tablets (ie, eCOA) at the site.














































#### CONFIDENTIAL

























#### 10.11. Fitzpatrick Skin Phototype

| Туре | Description |
|------|-------------------------------------------------------------|
| I | Always burns easily; never tans (sensitive) |
| II | Always burns easily; tans minimally (sensitive) |
| III | Burns moderately; tans gradually (light brown) (normal) |
| IV | Burns minimally; always tans well (moderate brown) (normal) |
| V | Rarely burns; tans profusely (dark brown) (insensitive) |
| VI | Never burns; deeply pigmented (insensitive) |

Source: Federal Register 1999







**Allergan** 



#### CONFIDENTIAL

